CLINICAL TRIAL: NCT01840085
Title: Open-Label Phase III Clinical Trial to Evaluate the Safety of 0.03% DSC127 Gel in Chronic Use for Treating Diabetic Foot Ulcers ("DFU")
Brief Title: Open-Label Study in Diabetic Foot Ulcers (DFU), to Evaluate Safety of 0.03% DSC127 Topical Gel in Chronic Use
Acronym: STRIDE 5
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSC127-2012-05
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic foot ulcer; plantar neuropathic ulcer; plantar neuroischemic ulcer; Wagner Grade 1 or Grade 2 DFU
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.03% DSC127 topical gel (Experimental)
  Interventions: Drug: 0.03% DSC127 topical gel

INTERVENTIONS:
Drug: 0.03% DSC127 topical gel

SUMMARY:
To evaluate the safety of topical 0.03% DSC127 Gel when used for one or more continuous treatment periods on a chronic Wagner Grade 1 or 2 foot ulcer(target ulcer) or multiple ulcers in diabetic subjects. The maximum duration of any treatment period is 24 weeks.

DETAILED DESCRIPTION:
All eligible subjects enrolled will begin daily Treatment with topical 0.03% DSC127 gel until complete wound closure (defined as skin re-epithelialization without drainage or dressing requirement) or 24 weeks, whichever occurs first.

If a patient has multiple ulcers on one foot, all may be treated, within the maximum of 24 weeks. If the ulcer does not heal, after a wash out period of 1 week, a new treatment period of up to 24 weeks may be initiated. Ulcer may be retreated if it recurs or if a new ulcer develops that meets study criteria.

For the entire duration of each treatment period the standard of care for DFU will be maintained.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ambulatory subjects who are at least 18 years of age at screening
2. Have at least one ulcer:

   1. chronic ( present >1month)
   2. Wagner Grade 1 or Grade 2 ulcer (i.e. Partial- or full- thickness and not involving bone, tendon or capsule (probing to tendon or capsule) and/or penetrating to tendon or capsule.)
   3. with no sign of infection or osteomyelitis, and
   4. is located below the malleolus.
3. Have an ABI > 0.7, or have a TcPO2 > 40 mm Hg or great toe systolic pressure > 50 mmHg to ensure healing potential.
4. Have Type I or Type II diabetes under metabolic control as confirmed by glycosylated hemoglobin (HbA1c) of ≤ 14%, obtained at enrollment or within 30 days prior to study enrollment.
5. Female subjects of child-bearing potential must have a negative pregnancy test at the time of enrollment and at the initiation of each study treatment period.
6. Female subjects of child-bearing potential must be willing to use a medically acceptable method of birth control, such as Essure®, hormonal contraception (oral pills, implantable device or skin patch), intrauterine device, tubal ligation, double barrier, or abstinence during the treatment periods of study participation.
7. Ability and willingness to understand and comply with study procedures and to give written informed consent prior to enrollment in the study or initiation of study procedures

Exclusion Criteria:

1. Has a known hypersensitivity to any of the study medication components.
2. Exposure to any investigational product within 30 days of entry into study.
3. Has active malignant disease of any kind (with the exception of basal cell carcinoma). A subject, who has had a malignant disease in the past, was treated and is currently disease-free, may be considered for study entry. Disease-free is defined as in remission for at least 5 years.
4. Chronic liver dysfunction evidenced by transaminase levels > 2.5 times higher than the upper level of normal on two occasions.
5. Has a history of additional risk factors for TdP (eg. heart failure, hypokalemia, family history of Long QT Syndrome) or taking medication which are known to prolong QT/QTc (Appendix G)
6. Receiving hemodialysis or chronic ambulatory peritoneal dialysis (CAPD) therapy.
7. Prior radiation therapy of the foot with the ulcer under study.
8. Current use of systemic corticosteroids or immunosuppressants within 8 weeks prior to enrollment into the study
9. Sickle-cell anemia, Raynaud's or other peripheral vascular disease.
10. Subjects receiving a biologic agent to include growth factors and skin equivalents (Regranex, Apligraft, or Dermagraft) in the 7 days prior to exposure to DSC127.
11. Subject who, in the opinion of the investigator, has uncontrolled hypertension
12. Subject has an ulcer which is determined to be clinically infected and requires antimicrobials or agents known to affect wound healing or has been taking systemic antibiotics for more than 7 days for any reason. (Subjects with infection at the initial visit of the Screening Period can be re-screened three weeks later after a single course of antibiotic therapy (occurring concurrently - within three weeks of the initial visit, the antibiotic treatment must have completed and some washout (7 days) must have elapsed); if after that time infection is still present, the subject will be excluded.)
13. Subjects who, in the opinion of the investigator, have clinically significant anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The proportion of all subjects reporting Adverse Events and Serious Adverse Events related to study treatment | 2.5yrs

OTHER OUTCOMES:
Changes from baseline in laboratory evaluations (clinically significant changes) | 2.5yrs
Proportion of all subjects treated and terminating prematurely due to adverse events related to study treatment. | 2.5yrs

CONTACTS AND LOCATIONS:
Overall Officials: John Caminis, MD, Study Director — Integra LifeSciences Corporation
Locations (21):
- United States (21):
  - WILMAX Clinical Research, Mobile, Alabama
  - Reliance Institute of Clinical Research, Chino, California
  - Roy O. Kroeker, DMP, Inc., Fresno, California
  - Limb Preservation Platform (LPP), Fresno, California
  - Foot and Ankle Clinic, Los Angeles, California
  - Center for Clinical Research, Inc., San Francisco, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - Orange County Research Center, Tustin, California
  - Advanced Research Institute of Miami, Homestead, Florida
  - UF Health Orthopaedic Surgery Clinic, Jacksonville, Florida
  - Phoenix Medical Research, LLC, Miami, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - GF Professional Research, Miami Lakes, Florida
  - Barry University Clinical Research, North Miami Beach, Florida
  - Professional Health Care of Pinellas, St. Petersburg, Florida
  - Eastern Carolina Foot & Ankle Specialists, Greenville, North Carolina
  - O'Malley Foot and Ankle, Wilmington, North Carolina
  - Martin Foot & Ankle, York, Pennsylvania
  - Carolina Musculoskeletal Institute, Aiken, South Carolina
  - Endeavor Clinical Trials, San Antonio, Texas
  - Professional Education and Research Institute, Roanoke, Virginia